CLINICAL TRIAL: NCT04982614
Title: A Multi-site, Open-label Non-inferiority Trial to Assess Immunogenicity of Two Doses of the Nonavalent Human Papillomavirus (HPV) Vaccine Among Children, Adolescents and Young Adults (9-26 Years) Living With HIV vs Three Doses of Nonavalent HPV Vaccine Among HIV Uninfected Young Women (15-26 Years) in Eswatini
Brief Title: HPV Vaccination in HIV Infected and HIV Uninfected Adolescents in Eswatini
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Jhpiego (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Elaine J. Abrams, MD, Professor of Pediatrics and Epidemiology, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAT6912; 7200AA19CA 00003 (Other Grant/Funding Number: USAID)
Record Dates: First submitted 2021-07-20; First posted 2021-07-29 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: HPV Infection; Hiv; HPV Vaccine
Keywords: HPV; Adolescents living with HIV; HPV immunogenicity; Vaccine adherence
MeSH Terms: conditions — Papillomavirus Infections; Acquired Immunodeficiency Syndrome | interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 2-dose regimen group (Experimental): Boys and girls (aged 9-14 years) and young women (aged 15-26 years) living with HIV will receive a two-dose regimen of the HPV vaccine at baseline (Month 0) and Month 6.
  Interventions: Biological: Gardasil ® 9
- 3-dose regimen group (SOC) (Active Comparator): HIV-uninfected young women (aged 15-26 years) will receive the standard of care three-dose regimen of the HPV vaccine at baseline (Month 0), Month 2 and Month 6.
  Interventions: Biological: Gardasil ® 9

INTERVENTIONS:
Biological: Gardasil ® 9 — GARDASIL 9 is a vaccine indicated in girls and women 9 through 45 years of age for the prevention of the following diseases: Cervical, vulvar, vaginal, and anal cancer, and Genital warts (condyloma acuminata) caused by Human Papillomavirus (HPV).
  0.5-mL suspension for intramuscular injection as a single-dose vial and prefilled syringe at the following regimen/schedule: 9 through 14 years - 2-dose at 0, 6 to 12 months OR 3-dose at 0, 2, 6 months 15 through 45 years - 3-dose at 0, 2, 6 months
  Other Names: Human Papillomavirus 9-valent Vaccine, Recombinant; 9vHPV vaccine

SUMMARY:
This is a multi-site, open-label non-inferiority study of the 9vHPV vaccine among a population of children, adolescents and young women living with HIV in Eswatini. This protocol seeks to assess immunogenicity of a two-dose 9vHPV vaccine regimen among girls and boys (9-14 years) and young women (15-26 years) living with HIV on antiretroviral therapy versus a three-dose 9vHPV vaccine regimen among HIV uninfected young women (15-26 years) in Eswatini. The secondary objectives include examining the safety profiles of the two-dose 9vHPV regimen in those living with HIV and the three-dose 9vHPV regimen in HIV-uninfected young women, as well as measuring the completion of the vaccination series among those living with HIV and those who are not infected with HIV.

DETAILED DESCRIPTION:
Cervical cancer remains a significant threat to public health worldwide and remains the leading cause of cancer-associated mortality in women in Sub Saharan Africa. Cervical cancer-associated morbidity and mortality is preventable through HPV vaccination, and screening and treatment of pre-cancerous lesions. To date, there is no nationwide HPV vaccination program in Eswatini and the country is not eligible for Global Alliance for Vaccines and Immunization (GAVI) procurement of HPV vaccines, and yet the triad of HIV, sexually transmitted infections (STI) and cervical cancer generates a severe disease burden warranting immediate introduction of this intervention. Given the global limitations in vaccine supply and the high cost for procurement, country programs, including in Eswatini, must optimize vaccine resources in order to maximize HPV vaccine coverage.

ELIGIBILITY:
Inclusion Criteria:

For people living with HIV receiving two-dose regimen:

* Females 9-26 years and males 9-14 years,
* Documented HIV infection,
* Aware of HIV+ status,
* Currently receiving antiretroviral treatment (ART) for HIV infection for at least six months,
* Living in Eswatini,
* For individuals 18+ years: able to provide informed consent,
* For individuals 15-17 years: able to provide informed assent,
* For individuals 9-14 years of age: able to provide informed assent AND accompanied by an adult caregiver who is able to give informed consent,
* Intending to remain in the vicinity of the study sites for the study period

For reference group of HIV-uninfected women receiving three-dose regimen:

* Females 15-26 years,
* Documented negative HIV test at baseline
* Living in Eswatini,
* Able to provide informed assent (15-17 years) or informed consent (18-26 years)
* Intending to remain in the vicinity of the study sites for the study period

Exclusion Criteria:

For all participants:

* Diagnosis of other immunosuppressive diseases or receipt of immunosuppressive medications,
* Diagnosis of other acute or chronic illness,
* Receipt of other vaccinations within 2-3 weeks before or after study vaccination,
* Receipt of blood-derived products within 6 months before or during the study,
* Previous receipt of an HPV vaccine,
* Currently pregnant,
* Known allergies to a vaccine component

Ages: 9 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1403 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Anti-HPV geometric mean antibody titers | Month 7 (4 weeks post Month 6 vaccine dose)
  Serum antibodies against HPV antigens (IgG, IFNg, TNF, IL2, CXCL10, granzyme, perforin, PTX3). Geometric mean titers will be summarized by treatment group, and the ratios of mean GMTs between treatment and control and their 95% confidence intervals calculated around point estimates.
Number of seroconversions | Month 7 (4 weeks post Month 6 vaccine dose)
  Number of participants who seroconvert, defined as having no HPV antibodies pre-vaccination, but detectable HPV antibodies at 4 weeks post month 6 vaccine dose

SECONDARY OUTCOMES:
Number of participants with serious adverse events (SAE) | Up to 6 months
  Number of participants who reported experiences of SAE. SAE is defined as those that experienced death, life-threatening conditions or hospitalizations.
Number of participants completing vaccination series | Up to 6 months
  Number of eligible participants completing the 2-dose or 3-dose regimens will be tallied.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Abrams, MD, Principal Investigator — Columbia University; Xolisile Dlamini, Principal Investigator — Ministry of Health Eswatini
Locations (5):
- Eswatini (5):
  - AHF Lamvelase, Manzini
  - AHF Manzini, Manzini
  - Raleigh Fitkin Memorial Hospital, Manzini
  - AHF Matsapha, Matsapha
  - Baylor College of Medicine - Bristol Myers-Squibb Children's Clinical Centre of Excellence, Mbabane

IPD SHARING:
Plan to Share IPD: No
Data sharing plan is still under development. The plan will follow all in-country requirements for research conducted in Eswatini.